CLINICAL TRIAL: NCT00591175
Title: A Randomized Clinical Trial Assessing Smoking Cessation Interventions In Dental Clinic Smokers
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: NYU College of Dentistry (Other)
Responsible Party: Sponsor
Other Study IDs: 01-117; NCT00070798 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salvia
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Standard Care
  Interventions: Behavioral: Standard Care only
- 2: Standard Care with Hygienist Counseling
  Interventions: Behavioral: Dental Hygienist provided counseling + Brief Questionnaire
- 3: Standard Care with Hygienist Counseling & Personalized Risk Communication
  Interventions: Behavioral: Dental Hygienist provided counseling with personalized risk communication + Brief Questionnaire

INTERVENTIONS:
Behavioral: Standard Care only — Dentist Provided Standard Care, 3-month follow-up assessment, Clinic visit salivary cotinine test, 12-month follow-up assessment, Clinic visit salivary cotinine test
  Groups: 1
Behavioral: Dental Hygienist provided counseling + Brief Questionnaire — Dental Hygienist provided + Brief Questionnaire, 3-month follow-up assessment,Clinic visit salivary cotinine test, 12-month follow-up, Clinic visit salivary cotinine test assessment
  Groups: 2
Behavioral: Dental Hygienist provided counseling with personalized risk communication + Brief Questionnaire — Dental Hygienist provided counseling with personalized risk communication + Brief Questionnaire, 3-month follow-up assessment, Clinic visit salivary cotinine test, 12-month follow-up assessment, Clinic visit salivary cotinine test
  Groups: 3

SUMMARY:
The goal of this study is to see if giving patients information about how smoking affects oral health will help them quit smoking. What we learn from this study will help researchers find new ways to help smokers.

ELIGIBILITY:
Inclusion Criteria:

* Patient seeking routine dental care at NYU College of Dentistry and meets medical clearance for routine care
* Active smokers (active smoking as self-reported regular use of at least 10 cigarettes per day)
* Able to provide a telephone number or collateral contact information where they can be reached over the subsequent 12 months
* Fluent in English or Spanish

Exclusion Criteria:

* History of mouth or throat cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smokers who are also patients at the NYU College of Dentistry
Sampling Method: Non-Probability Sample
Enrollment: 1072 (Actual)
Dates: Start 2001-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
efficacy of varied smoking cessation interventions | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org